CLINICAL TRIAL: NCT05489926
Title: A Study to Explore Pamiparib Treatment in Epithelial Ovarian Cancer After Prior PARP Inhibitor Exposure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jianqing Zhu, MD, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PamiAP
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — pamiparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pamiparib (Experimental)
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — Pamiparib, 60mg PO BID

SUMMARY:
The PamiAP will be a Phase II, single-arm, open label study to explore the efficacy and safety of Pamiparib treatment in patients with Epithelial Ovarian Cancer（EOC） who have had exposure to prior a PARP (poly(ADP-ribose)-polymerase) inhibitor

DETAILED DESCRIPTION:
The landscape for treatment of Epithelial Ovarian Cancer（EOC） is rapidly changing. With the release of data from numerous studies exploring the role of PARP (poly(ADP-ribose)-polymerase) inhibitor as maintenance and treatment, approval has expanded significantly in recent years. However, with the widespread exposure of PARP inhibitor in the patients, whether another PARP inhibitor can be reused in patients with PARP inhibitor resistance or disease progression. We have no data regarding the efficacy or safety of a PARP inhibitor retreatment in patients who have had exposure to prior a PARP inhibitor.

The objective of this study was to evaluate the efficacy and safety of Pamiparib in patients with EOC who had previously been treated with PARP inhibitor, and to explore the characteristics of patients who responded to PARP inhibitor again.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent;
2. Age ≥18;
3. Histologically diagnosed relapsed non-mucinous epithelial ovarian cancer (EOC) (including primary peritoneal and/or fallopian tube cancer), including platinum-sensitive and platinum-resistant patients, and the proportion of platinum-resistant patients was less than 40%
4. ≥2 previous lines of treatment
5. Patients must have received one prior PARP inhibitor therapy:

   1. Prior PARP inhibitor for maintenance treatment: the duration of prior PARP inhibitor exposure must have been ≥12 months following a first line of chemotherapy or ≥6 months following a second or subsequent line of chemotherapy
   2. Prior PARP inhibitor for treatment: the duration of prior PARP inhibitor exposure must have been ≥4 months
6. Patients must have lesions that can be measured according to RECIST v1.1 criteria;
7. Life expectancy ≥16 weeks;
8. Eastern United States Cancer Collaboration Group (ECOG) score 0-1;
9. Pregnant women must agree to effective contraception ≥120 days during the study period and after the last drug administration, and the results of serum pregnancy tests were negative 7 days ≤ before the first drug administration;
10. Patients must have adequate organ function as indicated by the following laboratory values:

    1. Hemoglobin ≥ 9 g/dL
    2. Absolute neutrophil count (ANC) ≥1.5 x 109/L
    3. Platelets ≥ 80 x 109/L
    4. Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
    5. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN
    6. Serum creatinine <1.5 x ULN

Exclusion Criteria:

1. Prior treatment with Pamiparib;
2. Patients who are candidates for surgery after disease progression;
3. Patients who have been treated with chemotherapy, biologic therapy, immunotherapy, investigational agent, anti-cancer Chinese medicine, or anti-cancer herbal remedies ≤ 14 days (or ≤5 half-lives, whichever is shorter) prior to starting study drug, or who have not adequately recovered from the side effects of such therapy;
4. Patients who have undergone major surgery/surgical therapy for any cause ≤ 4 weeks prior to starting study drug. Patients must have adequately recovered from the treatment and have a stable clinical condition before entering the study;
5. Patients who have undergone radiotherapy for any cause ≤ 14 days prior to starting study drug. Patients must have adequately recovered from the previous treatment and have a stable clinical condition before entering the study;
6. Untreated and/or active brain metastases; i. A scan to confirm the absence of brain metastases is not required ii. Patients with treated brain metastases must be off corticosteroids for ≥ 14 days and have no signs or symptoms of progressive brain metastases
7. Inability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation
8. Patients with any of the following cardiovascular criteria:

   i. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days prior to Day 1 ii. Evidence of symptomatic pulmonary embolismwithin 4 weeks prior to Day 1 iii. Acute myocardial infarction ≤ 6 months prior to Day 1 iv. Heart failure of New York Heart Association Classification III or IV (see Appendix 12) ≤ 6 months prior to Day 1 v. ≥ Grade 2 ventricular arrhythmia ≤ 6 months prior to Day 1 vi. Cerebrovascular accident ≤ 6 months prior to Day 1
9. Patients with other malignant cancer i. Except for surgically excised non-melanoma skin cancer, adequately treated carcinoma in situ of the cervix, adequately treated low-stage bladder cancer, ductal carcinoma in situ treated surgically with curative intent, or a malignancy diagnosed ≥ 5 years ago with no current evidence of disease and no therapy ≥ 5 years prior to Day 1
10. Diagnosis of myelodysplastic syndrome (MDS);
11. Known human immunodeficiency virus (HIV) infection, active viral hepatitis, or active tuberculosis;
12. Use ≤ 10 days (or ≤ 5 half-lives, whichever is shorter), prior to Day 1, or anticipated need for food or drugs known to be strong or moderate cytochrome P450 (CYP) 3A inhibitors or strong CYP3A inducers;
13. Pregnancy or nursing:

    i. Females of childbearing potential require a negative serum pregnancy test ≤ 7 days before Day 1.
14. Known history of intolerance to the excipients of the pamiparib capsule;
15. Previous complete gastric resection, chronic diarrhea, active inflammatory gastrointestinal disease, or any other disease-causing malabsorption syndrome.

    i. Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed.
16. Active bleeding disorder, including gastrointestinal bleeding, as evidenced by hematemesis, significant hemoptysis, or melena ≤ 6 months before Day 1;
17. Any illness that investigator thinks makes the patient unsuitable for entry into the study;
18. Unsolved acute effects of prior therapy of ≥ Grade 2 i. Except for AEs not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
CBR at 4 months | Up to approximately 18 months
  Clinical Benefit Rate (CBR) was defined as percentage of participants with confirmed best overall response of complete response (CR), partial response (PR), stable disease (SD) sustained for at least 4 months was assessed by investigators according to RECIST v1.1

SECONDARY OUTCOMES:
PFS | Up to approximately 18 months
  Progression-free Survival（PFS）, the time from the first dosing of the study drug until the first objective recording of disease progression or death from any cause, whichever occurred first
ORR | Up to approximately 18 months
  Overall Response Rate（ORR）, ORR of Pamiparib in patients with EOC were assessed by investigators according to RECIST v 1.1
DOR | Up to approximately 18 months
  Duration of Response（DOR）, refers to the time from the beginning of the first assessment of a tumor as CR or PR to the first assessment of PD or death from any cause were assessed by investigators according to RECIST v 1.1
AE | Up to approximately 21 months
  Adverse Event（AE）, an AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China